CLINICAL TRIAL: NCT03809377
Title: Multi-panel Coding and Non-coding Transcriptional Responses as an Indicator of Individualised Responses to Radiation Effects in Radiation Therapy Patients
Brief Title: Transcriptional Responses as an Indicator of Individualised Responses to Radiation Effects (RTGene 2)
Status: Active, not recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRAS258792
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood donation during radiotherapy: Participants will be asked to donate a blood sample at 5 time points during and after radiotherapy
  Interventions: Procedure: Blood donation during radiotherapy

INTERVENTIONS:
Procedure: Blood donation during radiotherapy — Participants will be asked to donate a blood sample at 5 time points during and after radiotherapy

SUMMARY:
Peripheral blood samples will be taken with informed consent from radiotherapy patients before and during treatment fractions for sarcoma, breast, lung, gut, genitourinary and head & neck tumours at The Royal Marsden. Candidate genes identified by PHE, Columbia and/or in the literature as being specific to radiation responses will be assessed, together with genes relevant to systemic inflammatory and immune responses, to identify transcriptional responses for a range of doses and exposures on an inter-individual basis. Data will be analysed using existing and new statistical tools focused on count data modelling. The intended outcome is identification of a radiation specific panel of genes to inform individual radiation responses and if the results are favourable, a large scale follow up to this project is expected.

DETAILED DESCRIPTION:
Biomarkers of radiation exposure are recognised to form an important component of the 'toolkit' for initial triage assessment of potentially exposed individuals in a mass casualty radiation accident or incident. Furthermore, radiation is an important medical tool and biomarkers can contribute to longer term assessment of radiation effects and public health risks. The gene expression assay has been gaining popularity as a sensitive biological marker of radiation exposure with the potential to be used for truly individualised dosimetry. The possibility for this assay to be used for a large scale mass-casualty scenario has been proposed and tested in a recent inter-comparison exercise. However, a fuller understanding of genetic factors that contribute to individual radiation risks is needed to inform tailored screening approaches - i.e. to identify a truly radiation specific panel of genetics responses for use as a transcriptional biomarker.

At Columbia University, research has shown that transcriptional effects have the potential to be used as individualised predictors of radiosensitivity to early and late effects. At Public Health England (PHE), recently established molecular counting nCounter technology allows direct counting of nucleic acid molecules (DNA, mRNA, miRNA and lncRNA) without the need for enzymatic reaction or amplification steps hence reducing time for data collection. This new gene expression analysis technique has been assessed for radiation biodosimetry applications with promising results. Furthermore, gene expression has shown a high degree of promise as a marker for late effects of radiation, for instance normal tissue reactions following curative radiotherapy for breast cancer.

In the earlier pilot RTGene study the investigators found genes that are consistently down-regulated and up-regulated towards the end of the radiotherapy treatment. The next stage of this work (RTGene 2) will be to validate the nCounter data for a small number of new genes consistently found in the top 6 of differentially expressed. Importantly, in an attempt to identify genes which are promising biomarkers of susceptibility to radiation-induced toxicity, expression levels will need to be compared with normal tissue reaction to IR, and combined with longer term radiation toxicity data to identify genes with the most pronounced expression level fluctuations during and after radiotherapy.

Peripheral blood samples will be taken with informed consent from radiotherapy patients before and during treatment fractions for sarcoma, breast, lung, gut, genitourinary and head & neck tumours at The Royal Marsden. Candidate genes identified by PHE, Columbia and/or in the literature as being specific to radiation responses will be assessed, together with genes relevant to systemic inflammatory and immune responses, to identify transcriptional responses for a range of doses and exposures on an inter-individual basis. Data will be analysed using existing and new statistical tools focused on count data modelling. The intended outcome is identification of a radiation specific panel of genes to inform individual radiation responses and if the results are favourable, a large scale follow up to this project is expected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Requirement for external beam radiotherapy (large-field RT, over at least 2 weeks) for sarcoma, breast, lung, gastrointestinal, head & neck or genitourinary tumours
* Written informed consent

Exclusion Criteria:

* Previous radiotherapy
* Concurrent chemotherapy/biological therapy or chemotherapy/biological therapy preceding radiotherapy by less than 4 weeks
* Concurrent hormone therapy or hormone therapy preceding radiotherapy by less than 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiotherapy for cancer
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Validation of new transcriptional techniques | 24 months after all participants have finished radiotherapy and donated blood samples
  Using nCounter platform to validate biomarkers of individual radiation exposure, in vivo

CONTACTS AND LOCATIONS:
Overall Officials: Navita Somaiah, Principal Investigator — The Institute of Cancer Research, London, UK
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided